CLINICAL TRIAL: NCT06418256
Title: Physiology and Pathologies Linked to Human Splenic Function : Direct and Ex-vivo Perfusion Explorations
Acronym: SPLEENVIVO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut Pasteur (Industry); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI17003; 2024-A00654-43 (Other: IDRCB Number)
Record Dates: First submitted 2024-05-13; First posted 2024-05-17 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Splenectomy
Keywords: Spleen; Human splenic physiology; Splenic clearance; Splenic filtration mechanisms; Perfusion experiments; Role of the spleen in the adaptive immune response; Genetic spleen mechanisms; Blood; Erythrocytes; Leukocytes; Lymphocytes; Malaria; Sickle cell disease; Hereditary spherocytosis
MeSH Terms: conditions — Malaria; Anemia, Sickle Cell; Spherocytosis, Hereditary | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Spleen fragments Peripheral blood cells Splenic blood cells, including red blood cells and Peripheral Blood Mononuclear Cells Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Adult patients cared in one of the APHP hospital (Necker-Enfants Malades Hospital, Saint-Antoine Hospital, Pitié Salpêtrière Hospital and Beaujon Hospital) for whom a splenic intervention (spleno-pancreectomy, or a total or partial splenectomy) is planned as part of their treatment.
  Interventions: Other: Spleen, blood and plasma collection

INTERVENTIONS:
Other: Spleen, blood and plasma collection — Adult patients for whom a splenic intervention (spleno-pancreectomy, or a total or partial splenectomy) is planned as part of their care. One or more tubes of venous blood collected for the care will be recovered following the pre- or intra-operative assessment. Immediately following surgery, after careful examination by the pathologist in charge, the whole spleen or spleen fragments will be collected for further analysis. Whenever possible a catheter will be introduced in the splenic artery, the spleen will be flushed/rinsed with 0.1 - 2 L of cold perfusion medium then transferred to the laboratory for ex-vivo perfusion. Before and at the end of the ex-vivo perfusion, splenic blood and spleen fragments will be collected and processed for further analyses.

SUMMARY:
Human splenic physiology remains poorly understood due to lack of functional exploration. However, through its ability to recognize alterations or modifications in circulating cells and to trigger an innate and adaptive response in response to these anomalies, the spleen plays a central role in several diseases affecting blood cells, directly or indirectly. The analysis of the splenic clearance of abnormal cells during ex-vivo perfusions made it possible to clarify the pathogenesis of malaria and the role of the spleen in the adaptive immune response. The study's investigative team wishes to extend these explorations to other human diseases in which the spleen is involved, and to evaluate the preventive or curative potential of substances that can modify the perception of blood cells by the spleen (e.g. monoclonal antibodies directed against circulating cells, among other options).

DETAILED DESCRIPTION:
Human splenic physiology remains poorly understood due to lack of functional exploration. However, through its ability to recognize alterations or modifications in circulating cells and to trigger an innate and adaptive response in response to these anomalies, the spleen plays a central role in several diseases affecting blood cells, directly or indirectly. The analysis of the splenic clearance of abnormal cells during ex-vivo perfusions made it possible to clarify the pathogenesis of malaria and the role of the spleen in the adaptive immune response. The study's investigative team wishes to extend these explorations to other human diseases in which the spleen is involved, and to evaluate the preventive or curative potential of substances that can modify the perception of blood cells by the spleen (e.g. monoclonal antibodies directed against circulating cells, among other options).

Participation to the study will be proposed to adult patients in whom a splenic intervention (spleno-pancreatectomy, or a total or partial splenectomy) is planned as part of their treatment.

One or more tubes of venous blood collected for the care will be retrieved following the pre- or intra-operative assessment. These samples will serve as controls during analyzes of splenic filtration mechanisms and/or perfusion experiments with populations of altered or modified cells and/or immunological and/or genetic analyses. Immediately following surgery, after careful examination by the pathologist in charge, the whole spleen or spleen fragments will be collected for further analysis. Whenever possible a catheter will be introduced in the splenic artery, the spleen will be flushed/rinsed with 0.1 - 2 L of cold perfusion medium then transferred to the laboratory for ex-vivo perfusion. Samples from different experimental conditions (for example red blood cell containing malaria parasite for a culture) may be introduced in the perfusion system pour kinetic analyses. Before and at the end of the ex-vivo perfusion, splenic blood and spleen fragments will be collected and processed for further analyses by cytology, cytometry, histology, immunohistochemistry, electronic microscopy, biochemistry, molecular biology, single cell analyses, on any other method. Peripheral and splenic blood samples or cells, as well as spleen fragments will be stored in. a biobank for further use or experimental analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patient requiring left splenopancreectomy or planned splenectomy regardless of the method or indication

Exclusion Criteria:

- The patient notified his doctor of his refusal to recover his spleen and blood volume

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with no age limit cared in one of the APHP hospital (Necker-Enfants Malades Hospital, Saint-Antoine Hospital, Pitié Salpêtrière Hospital and Beaujon Hospital) for whom a splenic intervention (spleno-pancreectomy, or a total or partial splenectomy) is planned as part of their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-10-16 (Actual); Primary Completion 2031-10-16 (Estimated); Study Completion 2031-10-16 (Estimated)

PRIMARY OUTCOMES:
Refine the understanding of spleen role during infections and conditions of the red blood cell and other human blood cells | Day 0
  Ability of the isolated-perfused human spleen to filter altered cell populations.

SECONDARY OUTCOMES:
Exploring splenic immunological mechanisms | Day 0
  Explore splenic immunological mechanisms including the maintenance of long-term memory against Plasmodium sp antigens. and other infectious agents: Bartonella sp., Babesia sp., smallpox virus, measles, hepatitis.
Kinetics of splenic clearance of altered or modified circulating elements | Day 0
  Explore the spleen filter role during infections, illnesses or use of blood cells, including properties of cells retained in the spleen, possibily after modification in vitro.
Exploring splenic clearance mechanisms | Day 0
  Clearance mechanisms: tissue and cellular topography and concentration of deposition of normal or altered or modified cells in the spleen (Histology, Imaging, Electron Microscopy, etc.).
Exploring the genetic control of spleen function | Day 0
  Genetic control of spleen function.
Explore the impact of preservation processes on organ and cell functions, as well as engraftment | Day 0
  Testing optimized freezing methods with evaluation of cell function in vitro and engraftment in a mouse model.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Buffet, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (5):
- France (5):
  - Hôpital Beaujon, Clichy
  - Hôpital Saint Antoine, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Institut Pasteur, Paris

IPD SHARING:
Plan to Share IPD: No